CLINICAL TRIAL: NCT05024799
Title: Effect of Different Sedation and Analgesia Strategies on Patients With Mechanical Ventilation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, JinyanXing, Director, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: QYFYKYLL931311920
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency | interventions — Fentanyl; Propofol; Butorphanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- F-P group (Experimental): the combination of fentanyl and propofol
  Interventions: Drug: Fentanyl, propofol
- F-D group (Experimental): the combination of fentanyl and dexmedetomidine
  Interventions: Drug: fentanyl and dexmedetomindine
- B-P group (Experimental): the combination of butorphanol and propofol
  Interventions: Drug: Butorphanol and propofol
- B-D group (Experimental): the combination of butorphanol and dexmedetomidine
  Interventions: Drug: Butorphanol and dexmedetomindine

INTERVENTIONS:
Drug: Fentanyl, propofol — The patients in this group will be administered with fentanyl and propofol
  Arms: F-P group
Drug: fentanyl and dexmedetomindine — The patients in this group will be administered with fentanyl and dexmedetomindine
  Arms: F-D group
Drug: Butorphanol and propofol — The patients in this group will be administered with butorphanol and propofol
  Arms: B-P group
Drug: Butorphanol and dexmedetomindine — The patients in this group will be administered with butorphanol and dexmedetomindine
  Arms: B-D group

SUMMARY:
Most patients in ICU are treated with a combination of analgesics and sedatives in most cases. Due to the different mechanism of different sedative and analgesic drugs, different antagonistic or synergistic effects may occur when combined with drugs, resulting in different clinical effects, especially significant effects on ventilators for patients with assisted breathing. Therefore, this study hopes to compare the effects of different sedative and analgesic drug combinations on the duration of mechanical ventilation for patients with ventilators, so as to guide the clinical adoption of a more reasonable sedative and analgesic scheme.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are treated with sedation and analgesia for invasive mechanical ventilation

Exclusion Criteria:

* they have baseline severe cognitive impairment; were pregnant or breast-feeding; were blind, deaf ; had second-degree or third-degree heart block or bradycardia requiring intervention; had an allergy to the experimental drugs; had an indication for benzodiazepines; were anticipated to have immediate discontinuation of mechanical ventilation; were expected to have neuromuscular blockade for more than 48 hours; were in a moribund state; or had received mechanical ventilation for more than 96 hours before meeting all inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
ventilator-free days at 28 days | at 28 days

IPD SHARING:
Plan to Share IPD: Undecided